CLINICAL TRIAL: NCT01137916
Title: Phase II Study to Evaluate Glivec (Imatinib Mesylate) to Induce Progression Arrest in Aggressive Fibromatosis / Desmoid Tumors Not Amenable to Surgical Resection With R0 Intent or Accompanied by Unacceptable Function Loss
Brief Title: Study to Evaluate Imatinib in Desmoid Tumors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Heidelberg University (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Bernd Kasper, PD Dr. med., Heidelberg University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSTI571BDE70
Record Dates: First submitted 2010-06-02; First posted 2010-06-07 (Estimated); Last update posted 2017-05-03 (Actual); Status verified 2017-05

CONDITIONS: Aggressive Fibromatosis; Desmoid Tumor
MeSH Terms: conditions — Desmoid Tumors | interventions — Imatinib Mesylate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- drug (Experimental): Imatinib 800 mg
  Interventions: Drug: Imatinib

INTERVENTIONS:
Drug: Imatinib — 800 mg
  Other Names: Glivec

SUMMARY:
The objective of the present study is to evaluate the activity and safety of imatinib in patients with aggressive fibromatosis who, after receiving the standard therapy, show an inoperable recurrent tumor or disease not readily controllable by surgery or radiotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histological confirmed aggressive fibromatosis (desmoid tumor)
* Measurable disease according to the RECIST criteria
* Evidence of relapse or disease progression within the last 6 months (based on RECIST criteria) in computed tomography or magnetic resonance imaging
* No possibility of complete surgical resection or cases in which surgical therapy leaving a large tissue defect, functional deficit or disfigurement would be required
* No possibility of curative radiotherapy with acceptable toxicity and/or late morbidity
* Previous treatment of the tumor region by surgical intervention and/or radiotherapy and/or antihormonal therapy possible
* Age > or = 18 years
* WHO PS < or = 1
* Effective contraception during study medication
* Signed informed consent form

Exclusion Criteria:

* Surgical intervention < 4 weeks
* Prior therapy with imatinib
* Pregnancy or lactation
* Severe hepatic dysfunction
* Known allergic reaction to imatinib or one of its components
* The following laboratory values: Absolute neutrophil count < 1.5 x 103/mm3, Platelets < 100,000/mm3, Serum creatinine > or = 2.5 mg/dl, SGOT and/or SGPT > 2.5 x ULN (upper limit of normal), Total bilirubin > 1.5 x ULN
* Participation in another study (four weeks before and during the study)
* Prior malignancy apart from completely resected basal cell carcinoma of the skin or carcinoma in situ of the uterine cervix

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2010-06; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Non-progression rate after 6 months of treatment | 6 months

SECONDARY OUTCOMES:
Non-progression rate after 12 and 24 months of treatment | 12 and 24 months
Response rate | 12 and 24 months
Progression-free survival (PFS) and overall survival (OS) | 12 and 24 months
Recording of patient quality of life | 12 and 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Bernd Kasper, PD Dr. med., Principal Investigator — University of Heidelberg, Mannheim University Medical Center
Locations (1):
- University of Heidelberg, Mannheim University Medical Center, Mannheim, Germany

REFERENCES:
- [Derived] Kasper B, Gruenwald V, Reichardt P, Bauer S, Rauch G, Limprecht R, Sommer M, Dimitrakopoulou-Strauss A, Pilz L, Haller F, Hohenberger P. Imatinib induces sustained progression arrest in RECIST progressive desmoid tumours: Final results of a phase II study of the German Interdisciplinary Sarcoma Group (GISG). Eur J Cancer. 2017 May;76:60-67. doi: 10.1016/j.ejca.2017.02.001. Epub 2017 Mar 8. PMID 28282612
- [Derived] Kasper B, Gruenwald V, Reichardt P, Bauer S, Hohenberger P, Haller F. Correlation of CTNNB1 Mutation Status with Progression Arrest Rate in RECIST Progressive Desmoid-Type Fibromatosis Treated with Imatinib: Translational Research Results from a Phase 2 Study of the German Interdisciplinary Sarcoma Group (GISG-01). Ann Surg Oncol. 2016 Jun;23(6):1924-7. doi: 10.1245/s10434-016-5132-4. Epub 2016 Feb 9. PMID 26861905
- See also: Related Info — http://www.gisg.de